CLINICAL TRIAL: NCT04779892
Title: The Study of Infliximab (CMAB008 and Remicade) in Healthy Subjects to Compare the PK and Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMAB008HV-I
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Intervention Model Description: Biological: CMAB008 Biological: Remicade
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAB008 (Experimental)
  Interventions: Drug: Infliximab
- Remicade (Active Comparator)
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — 100mg/vial

SUMMARY:
A phase 1, Randomized, Double-blind, Parallel group, Sing-dose study to compare the Pharmacokinetics and Safety of CMAB008 and Remicade in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject (male) between the ages of 18 and 45 years.
* Subject with a body weight of ≥50 kg and ≤ 80 kg and a BMI between 19.0~26.0 kg/m2 (both inclusive);
* Healthy as determined by pre-study medical history, physical examination, vital signs and 12-lead electrocardiogram;

Exclusion Criteria:

* Those who have surgered 4 weeks before signing the informed consent;
* Those with mental, respiratory, cardiovascular, digestive, urinary, reproductive, skeletal and motor, blood, endocrine, nervous and other system diseases, or those with any previous immune diseases;
* Those who have received any drug treatment (including prescription drugs, over-the-counter drugs, biological products, Traditional Chinese medicine, vitamins, dietary supplements, etc.) and health care products within 4 weeks before signing the informed consent;
* Those who accepted biological drugs within 6 months before signing the informed consent, or accepted the TNF monoconal antibody drugs;
* Any one of HIV antibody, HBsAg, HBeAg, HBcAg, HCV antibody and Treponema pallidum antibody is positive;
* Either T cell immunospot test (T-SPOT) or antinuclear antibody is positive;
* Those who have infected within 30 days before administration, or serious infection associated with hospitalisation and/or which required inrravenous antibiotics within 3 months before administration.
* Vaccinated within 30 months before signing the informed conset, or plan to vaccinate during the trail;
* Those who have used soft drugs within 3 months prior to signing the informed consent or hard drugs within 1 year prior to the trail; those who have positive drug abuse test results;
* Those who drinking too much tea, coffee and/or caffeinated beverages (more than 8 cups, 250ml per cup) every day;
* Those who have a blood donation history of 400 ml within 3 months, or 200 ml within 1 month;
* Those who have a history of drug or food allergy, or are known to be allergic to any component of the test drug or latex, etc.
* Those who are addicted to smoking or smoke more than 10 cigarettes per day on average within 6 months before signing the informed consent;
* Alcoholics or regular drinkers within 3 months before the trail, i.e. those who drink more than 14 units of alcohol per week (14 bottles of 360 ml beer or 630 ml spirits with 40% alcohol), or whose alcohol breath test is positive;
* Those who plan to donate sperm within 6 months after the adminstration of the test drug;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 1680 Hours After the Single Infusion of CMAB008/Remicade | up to 1680 hours

SECONDARY OUTCOMES:
Maximum Concentration of Infliximab After the Single Infusion of CMAB008/Remicade | up to 1680 hours
Time of Maximum Concentration of Infliximab After the Single Infusion of CMAB008/Remicade | up to 1680 hours
Area Under the Plasma Concentration-time Curve From Zero (0) Hours Extrapolated to infinite time After the Single Infusion of CMAB008/Remicade | up to 1680 hours
Total Frequency of AE/SAE Within the Whole Time of the Study | up to 1680 hours
Percentage of Patients in Whom Bind or Neutralizing Antibodies to Infliximab Were Detected | up to 1680 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Su Y, Li J, Wang C, Zhang X, Hou S, Guo H, Deng C, Ou L, Wang J. Population Pharmacokinetics of CMAB008 (an Infliximab Biosimilar) and Remicade(R) in Healthy Subjects and Patients with Moderately to Severely Active Rheumatoid Arthritis. Adv Ther. 2023 Mar;40(3):1005-1018. doi: 10.1007/s12325-022-02396-8. Epub 2023 Jan 6. PMID 36607544